CLINICAL TRIAL: NCT07081269
Title: Physical Fitness and Hot Executive Function in Alzheimer's Risk
Status: Recruiting | Type: Observational
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yu-Kai Chang, Principal Investigator, National Taiwan Normal University
Other Study IDs: PACNL_HPF_HEF
Record Dates: First submitted 2025-05-18; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Executive Function (Cognition); Event-Related Potentials; Physical Fitness
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults: Older adults, 50-70 years old.
  Interventions: Other: observation alone

INTERVENTIONS:
Other: observation alone — No interventions will be conducted during the observation period, maintaining participants' normal daily living conditions.
  Other Names: 1.5 year observation

SUMMARY:
This 18-month study tracks how physical fitness relates to executive function in older adults, aiming to determine if fitness improvements predict better cognitive performance. Participants complete assessments at baseline and 18 months, including cardiorespiratory fitness (YMCA bike test), muscle strength (chest and leg press tests), and executive function (computer tasks with brain activity recording via EEG). Additional measures include physical activity questionnaires, cognitive screening (MMSE), memory tests (digit span), demographics (age, sex, education), and blood tests for APOE ε4 gene status. No exercise program will be provided, allowing observation of natural fitness-cognition relationships in daily life.

DETAILED DESCRIPTION:
This prospective observational study examines associations between health-related physical fitness and behavioral/electrophysiological indices of cool and hot executive function in older adults over 18 months. The primary objective is to determine whether changes in physical fitness components predict concurrent changes in executive function domains.

Assessment Protocol: Participants complete comprehensive evaluations at baseline and 18-month follow-up, including: (1) cardiorespiratory fitness via YMCA submaximal cycle ergometry; (2) muscular strength through one-repetition maximum testing (chest press, leg press); and (3) executive function using computerized task-switching paradigms with simultaneous electroencephalography. Secondary measures include demographics (age, sex, education), physical activity levels (International Physical Activity Questionnaire-Taiwan Short Form), global cognition (Mini-Mental State Examination), and working memory (digit span forward/backward). Additionally, Apolipoprotein E ε4 (APOE ε4) genotype will be examined as a potential moderator of fitness-cognition relationships.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-70.
* Able to engage in fitness testing.
* Normal vision or corrected-to-normal vision.

Exclusion Criteria:

* Suffering from cardiopulmonary-related diseases.
* Suffering from cognitive, neurological or psychiatric disorders (e.g., dementia, Parkinson's disease, epilepsy, depression, schizophrenia, etc.).
* Suffering from infectious diseases (e.g., hepatitis, human immunodeficiency virus or Creutzfeldt-Jakob disease).
* Having a history of drug or alcohol abuse.
* Having colour vision deficiency (e.g., colour blindness).
* Having a family history of aneurysm.
* Taking medications that affect brain function.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is older adults aged 50-70.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in cardiorespiratory fitness | Approximately 25 minutes each at the baseline assessment and the 18-month follow-up post-assessment.
  Cardiorespiratory fitness will be estimated using the YMCA submaximal cycle ergometer test at baseline (Baseline Assessment) and at the 18-month follow-up (Post Assessment). Changes in cardiorespiratory fitness between the Baseline and Post Assessments will be evaluated.
Changes in muscular fitness | Approximately 25 minutes each at the baseline assessment and the 18-month follow-up post-assessment
  Muscular fitness will be assessed via a standardized 8-10 repetition maximum protocol on chest-press and leg-press machines at baseline (Baseline Assessment) and at the 18-month follow-up (Post Assessment). Changes in muscular fitness between the Baseline and Post Assessments will be evaluated.
Change in cognitive flexibility-response time | Approximately 30 minutes each at the baseline assessment and the 18-month follow-up post-assessment
  Cognitive flexibility will be assessed via a task-switching test at baseline (Baseline Assessment) and at the 18-month follow-up (Post Assessment). Changes in response times on the task-switching test between Baseline and Post Assessments will be analyzed.
Change in cognitive flexibility-adcuracy | Approximately 30 minutes each at the baseline assessment and the 18-month follow-up post-assessment
  Cognitive flexibility will be assessed via a task-switching test at baseline (Baseline Assessment) and at the 18-month follow-up (Post Assessment). Changes in accuracy on the task-switching test between Baseline and Post Assessments will be analyzed.
Change in EEG activity | Approximately 30 minutes each at the baseline assessment and the 18-month follow-up post-assessment
  Concurrent EEG data recorded during task switching at baseline (Baseline Assessment) and at the 18-month follow-up (Post Assessment) will be processed and analyzed. Differences in EEG activity between Baseline and Post Assessments will be examined.

SECONDARY OUTCOMES:
Cognitive function (Mini-Mental State Examination, MMSE) | Approximately 15 minutes each at the baseline assessment and the 18-month follow-up post-assessment
  The Mini-Mental State Examination (MMSE), a 30-item cognitive screening tool yielding a total score of 0-30, will be administered at baseline (Baseline Assessment) and at the 18-month follow-up (Post Assessment). Changes in MMSE total scores between Baseline and Post Assessments will be analyzed.
Working memory (Digit Span Tests) | Approximately 15 minutes each at the baseline assessment and the 18-month follow-up post-assessment
  Working memory will be assessed via the Digit Span subtest of the Wechsler Adult Intelligence Scale - Third Edition (WAIS-III), in which participants verbally reproduce auditorily presented digit sequences in their original (forward) or reverse (backward) order, at baseline (Baseline Assessment) and at the 18-month follow-up (Post Assessment). Changes in MMSE total scores between Baseline and Post Assessments will be analyzed.
ApoE genotype | 5 minutes at the Baseline Assessment
  Apolipoprotein E (ApoE) genotype will be determined for each participant by genotyping the single nucleotide polymorphisms rs429358 and rs7412.
Physical activity (Taiwan version of the International Physical Activity Questionnaire, IPAQ) | Approximately 15 minutes each at the baseline assessment and the 18-month follow-up post-assessment
  Physical activity will be assessed via the Taiwanese version of the International Physical Activity Questionnaire-Short Form (IPAQ-SF) at baseline (Baseline Assessment) and at the 18-month follow-up (Post Assessment). Changes in IPAQ-SF scores between Baseline and Post Assessments will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, PhD, Study Director — National Taiwan Normal University; Chine-Heng Chu, PhD, Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided